CLINICAL TRIAL: NCT07151794
Title: Correlation of G8, CARG, and Frailty Scales With Nutritional Biomarkers and G-CSF Requirement in Elderly Cancer Patients: A Prospective Study on Predicting Chemotherapy Toxicity
Brief Title: G8, CARG, Frailty, and Nutritional Markers in Predicting Chemotoxicity
Status: Active, not recruiting | Type: Observational
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Cemre Aydeğer, Research asistant, Çanakkale Onsekiz Mart University
Other Study IDs: COMU-FNO-2
Record Dates: First submitted 2025-07-31; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-01

CONDITIONS: Geriatric Oncology; Oncology; Nutrition; Nutrition Assessment
Keywords: G-CSF; CARG; Frailty; Mini Nutritional Assessment (MNA)
MeSH Terms: conditions — Neoplasms; Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: The study group consists of cancer patients aged 65 and older who are scheduled to receive at least two cycles of chemotherapy. Patients with hematological malignancies or receiving concurrent targeted, hormonal, immunotherapy, or radiotherapy are excluded.

SUMMARY:
This study aims to evaluate the ability of G8, CARG, and Frailty scales to predict chemotherapy-related toxicity and the need for G-CSF in elderly cancer patients. It also investigates their correlation with nutritional biomarkers (albumin, prealbumin, hemoglobin, CRP) and the Mini Nutritional Assessment (MNA) test.

DETAILED DESCRIPTION:
Background: Aging is associated with decreased physiological reserves, making elderly cancer patients more vulnerable to chemotherapy toxicity (CT). Traditional performance scales like ECOG may be insufficient for treatment decisions. Tools such as G8, Clinical Frailty Scale (CFS), and the Cancer and Aging Research Group (CARG) score are practical screening instruments recommended by ASCO and SIOG, yet their combined predictive accuracy for CT and granulocyte colony-stimulating factor (G-CSF) usage remains underexplored.

Objectives: This prospective study aims to evaluate the predictive performance of the G8, CARG, and Frailty scales-alone and in combination with nutritional biomarkers (albumin, prealbumin, hemoglobin, CRP)-in forecasting chemotherapy-related toxicity and G-CSF need. It also investigates the correlation between these geriatric assessment tools and Mini Nutritional Assessment (MNA) scores.

Methods: The study will be conducted at Çanakkale University Medical Faculty Oncology Outpatient Clinic. Patients aged 65 and above with a planned chemotherapy regimen will be recruited. Before the first chemotherapy cycle, patients will undergo G8, CARG, Frailty, and MNA assessments. Nutritional biomarkers will be extracted from pre-treatment routine lab tests. Chemotherapy toxicity and G-CSF requirement will be monitored across treatment cycles. ROC, correlation, and regression analyses will be conducted to evaluate predictive validity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Diagnosed with solid tumor malignancy
* Planned to undergo at least two cycles of adjuvant, neoadjuvant, or metastatic chemotherapy
* Clinically stable condition
* Provided written informed consent

Exclusion Criteria:

* Presence of hematological malignancies
* Concurrent hormonal therapy, targeted therapy, immunotherapy, or radiotherapy
* Acute infection or advanced organ failure (cardiac, hepatic, renal)
* Cognitive or psychiatric impairment preventing test participation
* Prior treatment with G-CSF

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study group consists of cancer patients aged 65 and older who are scheduled to receive at least two cycles of chemotherapy. Patients with hematological malignancies or receiving concurrent targeted, hormonal, immunotherapy, or radiotherapy are excluded.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Side effects of chemotherapy | From enrollment to 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Çanakkale Onsekiz Mart Univercity, Çanakkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bellera CA, Rainfray M, Mathoulin-Pelissier S, Mertens C, Delva F, Fonck M, Soubeyran PL. Screening older cancer patients: first evaluation of the G-8 geriatric screening tool. Ann Oncol. 2012 Aug;23(8):2166-2172. doi: 10.1093/annonc/mdr587. Epub 2012 Jan 16. PMID 22250183
- [Background] Church S, Rogers E, Rockwood K, Theou O. A scoping review of the Clinical Frailty Scale. BMC Geriatr. 2020 Oct 7;20(1):393. doi: 10.1186/s12877-020-01801-7. PMID 33028215
- [Background] Kenis, C., Bron, D., Libert, Y., et al., Relevance of a geriatric assessment in older patients with cancer: a systematic review, Journal of Geriatric Oncology, 2014, 5(2): 3-9.
- [Background] Decoster L, Van Puyvelde K, Mohile S, Wedding U, Basso U, Colloca G, Rostoft S, Overcash J, Wildiers H, Steer C, Kimmick G, Kanesvaran R, Luciani A, Terret C, Hurria A, Kenis C, Audisio R, Extermann M. Screening tools for multidimensional health problems warranting a geriatric assessment in older cancer patients: an update on SIOG recommendationsdagger. Ann Oncol. 2015 Feb;26(2):288-300. doi: 10.1093/annonc/mdu210. Epub 2014 Jun 16. PMID 24936581
- [Background] Wildiers, H., Heeren, P., Puts, M., et al., Comprehensive geriatric assessment (CGA) in older patients with cancer: facts and future, The Lancet Oncology, 2014, 15(5): e184-e192.
- [Background] Hurria A, Togawa K, Mohile SG, Owusu C, Klepin HD, Gross CP, Lichtman SM, Gajra A, Bhatia S, Katheria V, Klapper S, Hansen K, Ramani R, Lachs M, Wong FL, Tew WP. Predicting chemotherapy toxicity in older adults with cancer: a prospective multicenter study. J Clin Oncol. 2011 Sep 1;29(25):3457-65. doi: 10.1200/JCO.2011.34.7625. Epub 2011 Aug 1. PMID 21810685